CLINICAL TRIAL: NCT01160575
Title: A Semi-Factorial Cluster-Randomized Trial to Estimate the Effect Size of Community Mobilization and VCT Vans on the Adoption of Voluntary Counseling and Testing (VCT) Services in Andhra Pradesh, India: THE MCVCT STUDY
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910158; 10-I-N158
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-09-09

CONDITIONS: HIV; AIDS; Epidemiology; Prevention
Keywords: Counseling; Epidemiology; HIV; AIDS; Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
With an estimated 2.5 million HIV-infected persons, India is home to one of the largest populations of HIV-infected persons in the world. Yet, it is estimated that less than 20% of the people living with HIV in India are aware of their status. Andhra Pradesh (AP), situated in south India, is the state with the highest HIV burden in India. Reports from AP suggest usage of voluntary counseling and testing (VCT) is low, especially among high-risk groups. VCT has been shown to have many benefits in addition to diagnosis of HIV infection such as reduction in risk behavior, partner referral, and serving as an entry point to the health care system. Community mobilization and VCT vans have been shown in the past to play a role in increasing utilization of VCT services in various developing countries similar to India. The primary objective of this protocol is to arrive at an effect size of community mobilization alone, and both community mobilization and VCT vans, on the adoption of VCT services in Andhra Pradesh, India. Secondary objectives include identifying barriers to VCT, assessing stigma in the community, and establishing a specimen repository at the YRGCARE infectious disease laboratory in Chennai, India. We will achieve these objectives by conducting a cluster randomized clinical trial with 3 arms: ARM 1: standard of care with pre-existing VCT centers (SVCT); ARM 2: community mobilization in the setting of pre-existing VCT centers (CVCT); ARM 3: community mobilization plus VCT van in addition to the pre-existing VCT centers (MCVCT). The overall study duration will be 6 months from randomization. To our knowledge, this is the first study to examine the role of community mobilization and VCT vans on the adoption of VCT in the Indian context. It will provide us with vital data that will be used to plan a larger powered study to evaluate the effectiveness of these interventions including sites from other parts of India. Additionally, this study will also provide us with important information on barriers to VCT in these communities.

DETAILED DESCRIPTION:
With an estimated 2.5 million HIV-infected persons, India is home to one of the largest populations of HIV-infected persons in the world. Yet, it is estimated that less than 20% of the people living with HIV in India are aware of their status. Andhra Pradesh (AP), situated in south India, is the state with the highest HIV burden in India. Reports from AP suggest usage of voluntary counseling and testing (VCT) is low, especially among high-risk groups. VCT has been shown to have many benefits in addition to diagnosis of HIV infection such as reduction in risk behavior, partner referral, and serving as an entry point to the health care system. Community mobilization and VCT vans have been shown in the past to play a role in increasing utilization of VCT services in various developing countries similar to India. The primary objective of this protocol is to arrive at an effect size of community mobilization alone, and both community mobilization and VCT vans, on the adoption of VCT services in Andhra Pradesh, India. Secondary objectives include identifying barriers to VCT, assessing stigma in the community, and establishing a specimen repository at the YRGCARE infectious disease laboratory in Chennai, India. We will achieve these objectives by conducting a cluster randomized clinical trial with 3 arms: ARM 1: standard of care with pre-existing VCT centers (SVCT); ARM 2: community mobilization in the setting of pre-existing VCT centers (CVCT); ARM 3: community mobilization plus VCT van in addition to the pre-existing VCT centers (MCVCT). The overall study duration will be 6 months from randomization. To our knowledge, this is the first study to examine the role of community mobilization and VCT vans on the adoption of VCT in the Indian context. It will provide us with vital data that will be used to plan a larger powered study to evaluate the effectiveness of these interventions including sites from other parts of India. Additionally, this study will also provide us with important information on barriers to VCT in these communities.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Greater than or equal to 18 years of age
  2. Client to the clinic based standard VCT center or the VCT van during the study period
  3. Provides informed consent
  4. Must be a resident of the community for at least 6 months.
  5. Willing to complete survey
  6. Willing to provide a blood sample obtained by finger-stick or venipuncture for HIV testing.
  7. Willing to have blood samples stored.

EXCLUSION CRITERIA:

1. Participant is less than 18 years of age.
2. Study staff feels participant is psychologically unfit to understand the consent
3. Participant has already been enrolled in this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06-23; Study Completion 2014-09-09

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Quinn, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)

REFERENCES:
- [Background] Newmann S, Sarin P, Kumarasamy N, Amalraj E, Rogers M, Madhivanan P, Flanigan T, Cu-Uvin S, McGarvey S, Mayer K, Solomon S. Marriage, monogamy and HIV: a profile of HIV-infected women in south India. Int J STD AIDS. 2000 Apr;11(4):250-3. doi: 10.1258/0956462001915796. PMID 10772089
- [Background] Dandona L, Dandona R, Gutierrez JP, Kumar GA, McPherson S, Bertozzi SM; ASCI FPP Study Team. Sex behaviour of men who have sex with men and risk of HIV in Andhra Pradesh, India. AIDS. 2005 Mar 24;19(6):611-9. doi: 10.1097/01.aids.0000163938.01188.e4. PMID 15802980
- [Background] Simoes EA, Babu PG, John TJ, Nirmala S, Solomon S, Lakshminarayana CS, Quinn TC. Evidence for HTLV-III infection in prostitutes in Tamil Nadu (India). Indian J Med Res. 1987 Apr;85:335-8. PMID 3623641